CLINICAL TRIAL: NCT02063503
Title: The Identification of Prognostic Indicators for Exercise Therapy in Patients With Nonspecific Chronic Low Back Pain: A Multicenter Trial
Brief Title: Identification of Prognostic Indicators for Rehabilitation in Chronic Nonspecific Low Back Pain Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Denteneer Lenie, Dra. Denteneer Lenie, Universiteit Antwerpen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B300201215600
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Chronic Low Back Pain
Keywords: prognostic indicator; nonspecific; chronic; low back pain; Non specific chronic low back pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Low Back Pain | interventions — Physical Therapy Modalities; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Motor control therapy (Experimental): physiotherapy
  Interventions: Other: physiotherapy
- Isometric training therapy (Experimental): physiotherapy
  Interventions: Other: physiotherapy
- Combination therapy (Experimental): physiotherapy
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — every group receives 2 treatments every week during 9 consecutive weeks
  Other Names: - Motor control therapy; - Isometric training devices; - Combination therapy

SUMMARY:
There is a consensus that exercise therapy should be used as a therapy approach in CLBP but little consensus has been reached about the preferential type of therapy. There occurs to be a wash out effect because of the heterogeneous character of CLBP patients. As a result, no effect can be demonstrated for the entire sample. This is why one should consider creating subgroups based on prognostic indicators.

Objectives for this trial is to possibly identify prognostic indicators for treatment response to three forms of exercise therapy for patients with nonspecific chronic low back pain (CLBP).

The study design is a multicenter cohort design. Patients with nonspecific low back pain of more than three months duration are recruited in two different hospitals (Antwerp University Hospital and Sint Vincentius Hospital). After examination patients are assigned to one of three intervention groups: motor control therapy, isometric training therapy and a combination therapy. All patients will undergo eighteen treatment sessions during nine weeks. Measurements will be taken at baseline and after nine weeks of treatment.

The primary outcome used is the Modified Oswestry Disability Questionnaire (MDQ). For each type of exercise therapy prognostic indicators will be investigated.

Never before a multi-arm design was performed for the identification of prognostic indicators for exercise therapy in patients with nonspecific CLBP.

DETAILED DESCRIPTION:
Methods/ Design

Ethical approval (B300201215600) was obtained from the local ethics committees of the Antwerp University Hospital.

Study design In the identification of prognostic indicators is derived from a number of variables that have predictive potential for therapy outcome. These variables are obtained from baseline measurements and have a multidimensional character (impairments, activities/participation and contextual factors).

Patient recruitment Patients will be recruited by doctors at the service of two settings located in Antwerp namely the Antwerp University Hospital (UZA) and the Sint-Vincentius Hospital. Treatment and measurements will be performed at the site where the patient has been recruited.

Inclusion criteria: Current nonspecific LBP persisting at least three months, consulted a medical doctor during the last month because of the persistent low back pain, age between 18 and 60, sufficient fluency in Dutch to follow treatment instructions and answer survey questions.

Exclusion criteria: spinal canal stenosis, spondylolisthesis and spondylitis, large herniated disc sciatica, radiating pain below the knee, previous back surgery, a history of known spinal fractures, malignancy, known muscle-, nerve-, skin-, or joint diseases, pregnancy and lack of consent.

Measurements

Baseline testing As primary (dependent) outcome measure the Modified Oswestry Disability Questionnaire is used (MDQ). The MDQ is a disease specific questionnaire to measure disability in LBP patients [21-23].

As secondary (independent) outcome measures the following tests are used:

First, Measurement of impairments: duration of the LBP/ pelvis impairments / respiratory impairments (all three items through anamnesis). Prone instability test, Straight Leg Raise, Beighton scale, Active Straight Leg Raise, sitting knee extension test, waiters bow, pelvic tilt, side support test, extensor endurance test, active sit-up, Visual Analogue Scale for pain (VAS).

Second, measurement of limitations in activities and participation: hours of physical activity/week (trough anamnesis). Short Form 36 Health Survey (SF36), Roland Morris Disability Questionnaire (RMDQ).

Third, measurement of contextual factors: gender/ age / height / weight / body mass index / smoking / profession / underwent previous therapy / comorbidity (trough anamnesis). Tampa scale for kinesiophobia, Fear Avoidance Belief Questionnaire (FABQ), We performed a literature search to select all used clinical tests based on their reliability and validity [24]. The Baseline testing takes about 30 minutes.

Follow-up

Follow up takes place after completion of the treatment program at nine weeks. All patient reported outcome measures (PROMs) from the baseline testing will be re-evaluated at this moment.

Randomization & blinding

In the Sint-Vincentius Hospital, all included patients will follow the combination treatment since this is the only intervention group which is being organized in this hospital.

In the UZA, patients will be randomly assigned into one of the two treatment groups (motor control or isometric training) after baseline testing. The responsible researcher will use a randomization list generated with Microsoft ® Excel ® software (version 14.3.9, 2010 © Microsoft Corporation).

Intervention

During the nine weeks intervention, patients will be treated two times a week. Patients will be assigned randomly into one of three intervention groups (motor control therapy, isometric training therapy or combination therapy). Each intervention will take about seventy minutes. Ten minutes warming up and cooling down will be the same in each treatment regime. Each group receives fifty minutes of therapy specific intervention. Previously trained physiotherapists will give the treatment. To ensure that all therapists provide the same exercises, a treatment protocol for each treatment group was developed and a treatment diary will be filled out after each session.

Interventions in derivation and validation phase are similar.

Power analysis

This study describes the identification of prognostic indicators in which the therapeutic effect of the interventions cannot be predicted. Therefore, a two-tailed hypothesis was used to calculate the power. A pilot study showed that the standard deviation of the primary outcome measure, MDQ, is set at 10.53.6 Given these estimates, 54 patients were needed to detect a minimum clinically important difference (MCID, effect size 0.84) with 90% power. Consequently, three groups of 18 patients were needed to complete the trial.

Data analysis

Prognostic indicators aim to detect potential predictive variables for treatment success (dichotomous, yes/no) in a set of baseline measurements. A minimal decrease in the MDQ score of 9 points is considered as treatment success.

Potential predictive variables are selected as follows: first, individual variables from the self-reports, history, and physical examination are tested for their bivariate association with the reference standard using independent sample t tests, Mann-Whitney U tests or Chi-square tests based on the nature of the data. Variables with a significance level of P < 0.10 are retained as potential prediction variables. We choose a more liberal significance level at this stage to avoid excluding potential predictive variables.

This statistical analysis is performed for each treatment group (motor control therapy, general active exercise therapy and isometric training therapy).

Information form and informed consent

If patients meet the in- and exclusion criteria they are scheduled for an interview with one of our researchers to be informed about the trial. If patients decide to participate they will sign an informed consent. Information form and informed consent are made and have been approved by the ethics committee of the University of Antwerp.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 months low back pain
* consulted a medical doctor during last month because of persistent low back pain
* age between 18 - 60

Exclusion Criteria:

* vestibular dysfunction
* a history of known spinal fractures
* spondylolysis and spondylolisthesis
* radiating pain below the knee
* muscle, nerve, skin, joint diseases
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of functional disability | 2 years
  Modified Oswestry Low Back Pain Disability Questionnaire (MDQ): the patient questionnaire contains topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. Zero is equated with no disability and 100 being maximum disability.

SECONDARY OUTCOMES:
patient characteristics | 2 years
  gender (male/female), age (years), body height (cm), body weight (kg), hours of physical activity per week, duration of the LBP (months), sick leave (yes/no), smoking (yes/no), and pelvis impairments (yes/no)
clinical testing | 2 years
  Beighton scale (pos/neg), prone instability test (pos/neg), maximal range of motion of the straight leg raise (°), active straight leg raise (pos/neg), sitting knee extension test (pos/neg), waiters bow (pos/neg), pelvic tilt (pos/neg), side support test (seconds), extensor endurance test (seconds), active sit-up (pos/neg)
patient reported outcome measures | 2 years
  visual analogue scale for pain (score ranging 0-10), Roland Morris disability questionnaire (score ranging 0-24), Tampa scale for kinesiophobia (score ranging 17-68), short form 36 health survey (percentile) and the global perceived effect (score ranging 0-7)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Van Daele, Professor, Study Director — Universiteit Antwerpen; Gaetane Stassijns, Professor, Study Director — Universiteit Antwerpen, Universitair Ziekenhuis Antwerpen; Lenie Denteneer, phd student, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Denteneer L, Stassijns G, De Hertogh W, Truijen S, Jansen N, Van Daele U. Derivation and validation phase for the development of clinical prediction rules for rehabilitation in chronic nonspecific low back pain patients: study protocol for a randomized controlled trial. Trials. 2015 Jan 6;16:4. doi: 10.1186/1745-6215-16-4. PMID 25558975
- See also: official website of the University of Antwerp — http://www.uantwerp.be